CLINICAL TRIAL: NCT02991053
Title: Ultrasonography Guided Ilioinguinal /Iliohypogastric Block Versus Transversus Abdominis Plane Block in Intraoperative Anesthesia in Children - Randomized Controlled Study
Brief Title: Comparison of Transversus Abdominis Plane Block and Ilioinguinal / Iliohypogastric Nerve Block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Erzincan University (Other)
Responsible Party: Principal Investigator, ILKE KUPELI, assist. prof., Erzincan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ERZINCAN UNIVERSITY 8
Record Dates: First submitted 2016-12-04; First posted 2016-12-13 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-12

CONDITIONS: Intra-operative Anesthesia
Keywords: Intra-operative anesthesia; Pediatric patient; Transversus Abdominis Plane Block; ilioinguinal / iliohypogastric nerve block
MeSH Terms: interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- block and ketamine (Active Comparator): Transversus Abdominis Plane block after ketamine atropine induction and continued with ketamine only in anesthesia
  Interventions: Drug: ketamine
- block; ketamine with laryngeal mask; inhalation anesthesia (Active Comparator): After ketamine atropine induction, a laryngeal mask was inserted and anesthesia administration was continued with 2 sevoflurane minimum alveolar concentration and oxygen / air mixture and applied Transversus Abdominis Plane block.
  Interventions: Drug: ketamine
- block and ketamine ıh/ıl (Active Comparator): Ilioinguinal / iliohypogastric block after ketamine atropine induction and continued with ketamine only in anesthesia
  Interventions: Drug: ketamine
- ıh/ıl block; ketamine; inhalation anesthesia (Active Comparator): After ketamine atropine induction, a laryngeal mask was inserted and anesthesia administration was continued with 2 sevoflurane minimum alveolar concentration and oxygen / air mixture and applied Ilioinguinal / iliohypogastric block.
  Interventions: Drug: ketamine
- control group (Active Comparator): After ketamine atropine induction, a laryngeal mask was inserted and anesthesia administration was continued with 2 sevoflurane minimum alveolar concentration and oxygen / air mixture and Non-block, postoperative analgesia with paracetamol IV
  Interventions: Drug: ketamine

INTERVENTIONS:
Drug: ketamine

SUMMARY:
the aim of this study is to compare the effects of Transversus abdominis plane block and ilioinguinal / iliohypogastric block combined with sedation in pediatric surgeon on the anesthesia and analgesia contributions during surgery without general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* American society of anesthesia score I-II
* To undergo elective lower abdominal surgery
* between 2-6 years old

Exclusion Criteria:

* Patients with psychiatric disease
* Patients whose weight is more than 40 kg
* Patients with cardiac-pulmonary-neurological disease
* Patients with bleeding disorder
* Patients with infection or scar on the injection area
* Patients with known allergies to local anesthetics

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-08 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Amount of anesthetic drug which was used | 2 hour

SECONDARY OUTCOMES:
Postoperative visual analogue scale | one day

CONTACTS AND LOCATIONS:
Overall Officials: ilke kupeli, Principal Investigator — Erzincan University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Newman K, Ponsky T, Kittle K, Dyk L, Throop C, Gieseker K, Sills M, Gilbert J. Appendicitis 2000: variability in practice, outcomes, and resource utilization at thirty pediatric hospitals. J Pediatr Surg. 2003 Mar;38(3):372-9; discussion 372-9. doi: 10.1053/jpsu.2003.50111. PMID 12632352
- [Background] Scott AD, Phillips A, White JB, Stow PJ. Analgesia following inguinal herniotomy or orchidopexy in children: a comparison of caudal and regional blockade. J R Coll Surg Edinb. 1989 Jun;34(3):143-5. PMID 2810163
- [Background] Markham SJ, Tomlinson J, Hain WR. Ilioinguinal nerve block in children. A comparison with caudal block for intra and postoperative analgesia. Anaesthesia. 1986 Nov;41(11):1098-103. doi: 10.1111/j.1365-2044.1986.tb12956.x. PMID 3789367
- [Background] Tanaka M, Mori N, Murakami W, Tanaka N, Oku K, Hiramatsu R, Nakagawa M, Yasumoto K. [The effect of transversus abdominis plane block for pediatric patients receiving bone graft to the alveolar cleft]. Masui. 2010 Sep;59(9):1185-9. Japanese. PMID 20857679
- [Background] Stuart-Smith K. Hemiarthroplasty performed under transversus abdominis plane block in a patient with severe cardiorespiratory disease. Anaesthesia. 2013 Apr;68(4):417-20. doi: 10.1111/anae.12108. Epub 2012 Dec 17. PMID 23252578
- [Background] Tekelioglu UY, Demirhan A, Sit M, Kurt AD, Bilgi M, Kocoglu H. Colostomy with Transversus Abdominis Plane Block. Turk J Anaesthesiol Reanim. 2015 Dec;43(6):424-6. doi: 10.5152/TJAR.2015.89410. Epub 2015 Dec 1. PMID 27366540
- [Background] Polaner DM, Taenzer AH, Walker BJ, Bosenberg A, Krane EJ, Suresh S, Wolf C, Martin LD. Pediatric Regional Anesthesia Network (PRAN): a multi-institutional study of the use and incidence of complications of pediatric regional anesthesia. Anesth Analg. 2012 Dec;115(6):1353-64. doi: 10.1213/ANE.0b013e31825d9f4b. Epub 2012 Jun 13. PMID 22696610